CLINICAL TRIAL: NCT05673785
Title: A Phase 2, Single-Arm, Open-Label, Multicenter Study of Brentuximab Vedotin in Combination With Cyclophosphamide, Doxorubicin (Hydroxydaunorubicin), Prednisone (CHP) in the Frontline Treatment of Chinese Patients With CD30-Positive (CD30+) Peripheral T-Cell Lymphomas (PTCL)
Brief Title: A Study of Brentuximab Vedotin in Combination With Cyclophosphamide, Doxorubicin (Hydroxydaunorubicin), Prednisone (CHP) in Chinese Participants With CD30-Positive (CD30+) Peripheral T-Cell Lymphomas (PTCL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25024
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma | interventions — Brentuximab Vedotin; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin + CHP (Experimental): Brentuximab vedotin 1.8 mg/kg, intravenous (IV) infusion, within 1 hour of completing treatment with other IV agents, i.e., cyclophosphamide 750 mg/m^2 and doxorubicin 50 mg/m^2 IV, on Day 1 of each 21-day cycle, and prednisone 100 mg tablets, orally, on Days 1 through Day 5, for up to 8 cycles (6 months) or until progressive disease (PD), unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Brentuximab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin IV infusion
Drug: Cyclophosphamide — Cyclophosphamide IV infusion
Drug: Doxorubicin — Doxorubicin IV infusion
Drug: Prednisone — Prednisone tablets

SUMMARY:
This study will use a combination of Brentuximab vedotin with CHP to treat adult Chinese participants with CD30+ PTCL.

The main aims of the study are to evaluate:

* Side effect from the A+CHP
* Check how much A+CHP stays in their blood over time. This will help Takeda to work out the best dose to give people in the future.
* If A+CHP improves outcome of newly diagnosed CD30+ PTCL

Brentuximab vedotin will be given through vein on Day 1 of each 21-day cycle. Cyclophosphamide and doxorubicin will be given through vein. Prednisone will be given orally daily on Days 1 through 5.

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin. Brentuximab vedotin is being tested to treat CD30+ PTCL in Chinese participants. This study will look at the efficacy, safety, and pharmacokinetics (PK) of A+CHP as frontline treatment for newly diagnosed CD30+ PTCL.

The study will enroll approximately 52 participants. Participants will be enrolled in a single group to receive:

• Brentuximab vedotin 1.8 milligrams per kilogram (mg/kg) + Cyclophosphamide 750 milligrams per square meter (mg/m^2), Doxorubicin 50 mg/m^2 and Prednisone 100 mg

This multi-center trial will be conducted in China. The overall time to participate in this study is approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have newly diagnosed CD30+ PTCL, per the Revised European American Lymphoma 2016 World Health Organization (WHO) classification, by local assessment. Tumor specimen must be submitted before enrollment for subsequent central pathology review to confirm histology (and anaplastic lymphoma kinase (ALK) status, if applicable), and CD30 expression. Eligible histologies include:

   1. ALK-positive systemic anaplastic large cell lymphoma (sALCL) with an International Prognostic Index (IPI) score of ≥2.
   2. ALK-negative sALCL.
   3. PTCL- not otherwise specified (NOS).
   4. Angioimmunoblastic T-cell lymphoma (AITL).
   5. Enteropathy associated T-cell lymphoma (EATL).
   6. Hepatosplenic T-cell lymphoma (HSTCL).
2. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
3. Fluorodeoxyglucose (FDG)-avid disease by positron emission tomography (PET) imaging and measurable disease with at least 1 bidimensionally measurable lesion (>1.5 cm in its largest dimension) by computed tomography (CT).
4. Suitable venous access for the study-required blood sampling, including pharmacokinetic (PK) and immunogenicity sampling.
5. Clinical laboratory values as specified below at screening/baseline within 7 days before the first dose of study drug:

   1. Total bilirubin must be ≤1.5 times the upper limit of normal (ULN) or ≤3 times the ULN for participants with Gilbert's disease or documented hepatic involvement with lymphoma.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be ≤3 times the ULN or ≤5 times the ULN for participants with an elevation that can be reasonably ascribed to the presence of metastatic disease in liver.
   3. Serum creatinine must be <2.0 milligram per deciliter (mg/dL) and/or creatinine clearance or calculated creatinine clearance >40 milliliter (mL)/minute.
   4. Hemoglobin must be ≥8 grams per deciliter (g/dL). (Red blood cell transfusion is allowed ≥14 days before assessment.)
   5. Absolute neutrophil count >1.5×10^9/liter (L).
   6. Platelet count ≥75×10^9/L (unless documented bone marrow involvement with lymphoma).

Exclusion Criteria:

1. Systemic anticancer therapy, including traditional Chinese medicine with antitumor indication for disease under study before the first dose of study drugs.
2. Major surgery within 28 days before the first dose of study drug.
3. Known human immunodeficiency virus (HIV)-positive status.
4. Known hepatitis B virus (HBV) surface antigen (HBsAg) seropositivity or active hepatitis C virus infection.

   Note: Participants who have positive HBV core antibody and are HBsAg negative can be enrolled, but must have an undetectable HBV viral load.
5. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
6. Any of the following cardiovascular conditions or values within 6 months before the first dose of study drug:

   1. Left-ventricular ejection fraction <45%.
   2. Myocardial infarction within 6 months of enrollment.
   3. New York Heart Association Class III or IV heart failure.
7. Participants with current diagnosis of primary cutaneous CD30+ T-cell lymphoproliferative disorders and lymphomas. Participants with cutaneous anaplastic large cell lymphoma (ALCL) with extracutaneous tumor spread beyond locoregional lymph nodes are eligible (previous single-agent treatment to address cutaneous and locoregional disease is permissible).
8. Participants with mycosis fungoides (MF) [including transformed MF].
9. Uncontrolled diabetes mellitus.
10. Baseline peripheral neuropathy ≥Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE], version 5.0).
11. History of progressive multifocal leukoencephalopathy (PML).
12. Previous treatment with brentuximab vedotin or CD30 monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by Independent Review Facility (IRF) Assessment per Revised Response Criteria for Malignant Lymphoma | Up to approximately 7 months
  ORR by IRF assessment following the completion of study treatment is defined as the percentage of participants who have achieved a complete response (CR) or partial response (PR) by IRF assessment using the International Working Group (IWG) Revised Response criteria following the completion of study treatment. CR is defined as disappearance of all evidence of disease. PR is defined as regression of measurable disease and no new sites.
Percentage of Participants who Experience at Least One Treatment Emergent Adverse Event (TEAE) | Up to approximately 7 months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event that occurs after administration of the first dose of study treatment and up through 30 days after the last dose of study treatment.
Percentage of Participants With Clinically Significant Laboratory Test Values | Up to approximately 7 months
  Clinical laboratory tests will include hematocrit, hemoglobin, platelet (count), white blood cell (WBC) count, absolute neutrophil count (ANC), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (total), albumin, alkaline phosphatase, blood urea nitrogen, calcium, chloride, gamma glutamyl transferase, glucose, lactate dehydrogenase, phosphate, potassium, sodium, urate and creatinine evaluations. Any value outside the normal range will be flagged for the attention of the investigator who will assess whether or not a flagged value is of clinical significance.
Percentage of Participants With Clinically Significant Vital Signs | Up to approximately 7 months
  Vital signs will include measurements of diastolic and systolic blood pressure, heart rate, and body temperature. Any value outside the normal range will be flagged for the attention of the investigator who will assess whether or not a flagged value is of clinical significance.

SECONDARY OUTCOMES:
CR Rate by IRF Assessment per Revised Response Criteria for Malignant Lymphoma | Up to approximately 7 months
  CR rate by IRF assessment following the completion of study treatment is defined as the proportion of participants who have achieved a CR by IRF assessment using the IWG Revised Response criteria following the completion of study treatment. CR is defined as disappearance of all evidence of disease.
1-Year Progression Free Survival (PFS) Rate by IRF Assessment per Revised Response Criteria for Malignant Lymphoma | Up to approximately 12 months
  The 1-year PFS rate by IRF assessment using the IWG Revised Response criteria is defined as the percentage of participants alive and progression free at 1 year. PFS is defined as the time from the start of study treatment to the date of first documentation of PD, death due to any cause, or receipt of subsequent anticancer therapy to treat residual or PD, whichever occurs first.
1-Year Overall Survival (OS) Rate | Up to approximately 12 months
  The 1-year OS rate is defined as the percentage of participants alive at 1 year. OS is defined as the time from the start of study treatment to the date of death due to any cause.
ORR by IRF and Investigator Assessment per 2014 Lugano Classification | Up to approximately 7 months
  ORR by IRF and investigator assessment per 2014 Lugano Classification, assessed by integrated computed tomography (CT) and positron emission tomography (PET)-based responses are defined as the percentage of participants who have achieved a complete response (CR) or partial response (PR) by IRF and investigator assessment following the completion of study treatment.
CR Rate by IRF and Investigator Assessment per 2014 Lugano Classification | Up to approximately 7 months
  CR rate by IRF and investigator assessment per 2014 Lugano Classification, assessed by integrated CT and PET-based responses is defined as the percentage of participants who have achieved a CR by IRF and investigator assessment following the completion of study treatment.
Time to Response (TTR) by IRF and Investigator Assessment per 2014 Lugano Classification | Up to approximately 7 months
  TTR by IRF and investigator assessment per 2014 Lugano Classification, assessed by integrated CT and PET-based responses=time from date of first study drug administration to date of first documented objective response(CR or PR) by IRF and investigator assessment following the completion of study treatment for responders.
1-Year PFS Rate by IRF and Investigator Assessment per 2014 Lugano Classification | Up to approximately 12 months
  The 1-year PFS rate by IRF and investigator assessment per 2014 Lugano Classification is defined as the percentage of participants alive and progression free at 1 year. PFS is defined as the time from the start of study treatment to the date of first documentation of PD, death due to any cause, or receipt of subsequent anticancer therapy to treat residual or PD, whichever occurs first.
Duration of Response (DOR) by Investigator Assessment per 2014 Lugano Classification | Up to approximately 36 months
  DOR by investigator assessment using the 2014 Lugano Classification criteria is defined as the time between the first documentation of objective tumor response (CR or PR) by investigator assessment and the first subsequent documentation of objective tumor progression, death due to any cause, or receipt of subsequent anticancer therapy to treat residual or PD, whichever occurs first.
Serum Antibody-drug Conjugate (ADC) Concentration | Preinfusion and at multiple time points (Up to 96 hours [Cycle 1]/168 hours [Cycle 2]) postinfusion; Preinfusion up to Cycle 8, each cycle = 21 days
Plasma Monomethyl Auristatin E (MMAE) Concentration | Preinfusion and at multiple time points (Up to 96 hours [Cycle 1]/168 hours [Cycle 2]) postinfusion; Preinfusion up to Cycle 8, each cycle = 21 days
Percentage of Participants who are Antidrug Antibodies (ADA) Negative, ADA Transiently and Persistently Positive, ADA Titer, and Neutralizing Antidrug Antibody (Nab) Negative and Positive | Preinfusion on Day 1 of each cycle up to Cycle 8, each cycle = 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (16):
- China (16):
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial Peoples Hospital, Guangzhou
  - The First Affiliated Hospital of Zhejiang University school of medicine, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/a688e46576ec4dff?idFilter=%5B%22C25024%22%5D